CLINICAL TRIAL: NCT04041388
Title: Is Maxillary Segment Tipping During Transpalatal Distraction Related to the Vertical Level of the Horizontal Corticotomies and the Vertical Position of the Distractor Related to Dental and Bony Reference Planes?
Brief Title: Maxillary Segment Tipping During Transpalatal Distraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Veerle Van Mossevelde, Study Coordinator, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPD Studie v 1.0
Record Dates: First submitted 2019-07-31; First posted 2019-08-01 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Maxillary Hypoplasia
Keywords: Transpalatal; Maxillary expansion; Tooth-borne; Bone-borne; Distractor; Tipping; Osteotomy height
MeSH Terms: conditions — Retrognathia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tooth tipping (Other)
  Interventions: Other: Conebeam CT

INTERVENTIONS:
Other: Conebeam CT — medical imaging technique consisting of X-ray computed tomography where the X-rays are divergent, forming a cone

SUMMARY:
The investigator proposes a multi-centre study to investigate tipping of teeth, bringing into consideration the height of the osteotomy line and the height and placement of the transpalatal distractor as possible factors. If tipping occurs depending on these factors, the investigator could identify the situations that cannot be straightened by the orthodontist and provide another course of action for these specific patients.

DETAILED DESCRIPTION:
Surgically Assisted Rapid Maxillary Expansion (SARME) is widely accepted for the treatment of maxillary hypoplasia. The differences between SARME with a tooth-borne or a bone-borne distractor have already been extensively investigated, bringing to light that a bone-borne distractor has less negative side effects. One of the major concerns with the tooth-borne distractor is the tipping of the anchor teeth, which is bypassed by the bone-borne distractor which applies its force directly on the bone. One study investigated the tipping of teeth with a bone-borne distractor in 10 patients, showing that there was a minor change in the tooth axis. The investigator proposes a multi-center study to investigate this tipping further, bringing into consideration the height of the osteotomy line and the height and placement of the transpalatal distractor as possible factors. If tipping occurs depending on these factors, the investigator could identify the situations that cannot be straightened by the orthodontist and provide another course of action for these specific patients.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing a surgically assisted rapid maxillary expansion with a bone borne transpalatal distractor.
* Cone beam CT pre op and 3 weeks post op is available

Exclusion Criteria:

* Complication of the process by e.g. surgical site infection
* Asymmetrical expansion of more than 3.0 mm measured at the central incisivae occurred

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Tooth axis | 3 weeks postoperatively
  To investigate changes in the tooth axis of the first and second (pre-)molars bilaterally in the upper jaw before and after surgically assisted rapid maxillary expansion using a bone borne transpalatal distractor.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Van Bogaert, MD, Principal Investigator — Universitair Ziekenhuis Brussel; Maurice Mommaerts, Prof MULT, Study Director — Universitair Ziekenhuis Brussel; Nathalie Loomans, MD, Study Chair — GasthuisZusters Antwerpen (GZA); Yannick Spaey, MD, Study Chair — Mariaziekenhuis Noord-Limburg
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Vlaams Brabant, Belgium